CLINICAL TRIAL: NCT00583518
Title: Open Label, Multi-centre, Longitudinal, Prospective, Phase IV Clinical Trial to Compare Two Image Technologies (ImaTx and DXA) Assessing the Anabolic Effects of PTH(1-84) in Postmenopausal Women With Primary Osteoporosis
Brief Title: STEP: Study of Imaging Techniques (ImaTx and DXA) in Postmenopausal Women With OstEoporosis Using Preotact (FP-008-ES)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP-008-ES
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2012-05-07 (Estimated); Status verified 2012-05

CONDITIONS: Postmenopausal Women With Primary Osteoporosis
MeSH Terms: interventions — Parathyroid Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Parathyroid hormone (PTH) — Postmenopausal women with primary osteoporosis
  Other Names: Preotact

SUMMARY:
The primary objective of the study is to explore the relationship between a new image technology (ImaTx), that analyzes the trabecular structure of the bone using digitized radiographs and the bone mineral density (BMD) measured by Dual X-ray Absorptiometry (DXA) in the lumbar spine of postmenopausal (PM) women with osteoporosis (OP) after treatment with PTH (1-84).

ELIGIBILITY:
Inclusion Criteria:

1. Has the subject given informed consent according to local requirements before any trial-related activities? A trial-related activity is any procedure that would not have been performed during the routine management of the subject.
2. Is the subject a female?
3. Is the subject 65 years old or above?
4. Is the subject postmenopausal (more than 5 years), in the judgement of the investigator?
5. Does the subject have primary osteoporosis, with a lumbar spine T score ≤ -3.0 SD, or a lumbar spine T-score ≤ -2.5 SD and previous fragility fracture[1], with a minimum of two evaluable lumbar vertebrae?
6. Does the subject have a life expectancy of > 2 years?
7. Does the subject have a clinical indication to receive PTH(1-84) and is able to self-inject (or to have PTH(1-84) injection by a helper)?

All inclusion criteria must be answered "yes" for a subject to participate in the trial.

[1] Definition of fragility fracture in the scope of the study: Bone fractures that occur as a result of a fall from standing height or less. That is, fractures resulting from mechanical forces that would not ordinarily cause fractures in a healthy person.

Exclusion Criteria:

1. Is the patient currently taking any of the following treatments: bisphosphonates, selective estrogen receptor modulators or hormone replacement therapy (if the patient discontinues any of these treatments at the screening visit, the question can be answered NO and the patient can be included)?
2. Has the subject received, during her lifetime, strontium, fluoride or calcitonin > 3 months in total?
3. Has the subject ever been treated with teriparatide or PTH(1-84)?
4. Is the subject taking any other medication known to affect bone metabolism in the opinion of the investigator?
5. Has the subject ever received radiation therapy to the skeleton?
6. Has the subject ever been treated for a bone malignant disease?
7. Is the subject suffering from any known clinically significant diseases affecting calcium metabolism, including metabolic bone diseases such as hyperparathyroidism, Paget's disease, osteogenesis imperfecta, or osteomalacia?
8. Does the subject have any known history of hypersensitivity to parathyroid hormone or any of the excipients in the drug?
9. Does the subject have an elevated serum calcium (total serum calcium value >10.2 mg/dl) after at least 14 days of a 1000 mg calcium and 800 IU vitamin D3 supplementation?
10. Does the subject have a clinically significant elevation of serum alkaline phosphatase judged by the investigator?
11. Does the subject have an impaired kidney function with creatinine clearance <30ml/min (indirect measurement by serum creatinine)?
12. Does the subject have a severe hepatic impairment, defined as > 9 Child-Pugh score?
13. Has the subject participated in a clinical trial with an Investigational Medicinal Product (IMP) during the last 30 days?
14. Does the subject have a bilateral hip replacement?

All exclusion criteria must be answered "no" for a subject to participate in the trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2007-11; Primary Completion 2011-11 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient between the percentage of increase in Bone Mineral Density (BMD) obtained by DXA in the lumbar spine and in Trabecular Fragment Length (TFL) obtained by ImaTx in digitised radiographs of lumbar spine from baseline to EOT | 72 weeks

SECONDARY OUTCOMES:
BMD obtained by DXA in the lumbar spine (DXA SPI BMD). Two measurements will be determined: Mean value (g/cm2) and percentage of increase at EOT versus baseline (%). | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark